CLINICAL TRIAL: NCT04055675
Title: The Frequency of Leukocytes and Nitrites in the Urine of Healthy Adults
Brief Title: Urinalysis Results in Healthy Individuals
Status: Completed | Type: Observational
Sponsor: Kendall Healthcare Group, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-356 Non-NSU Health
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Results first posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Asymptomatic Bacteriuria; Asymptomatic Pyuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asymptomatic Male Volunteers: These are subjects over the age of 18 who have no acute symptoms, volunteered to provide a urine sample, and are male.
  Interventions: Diagnostic Test: Urine dipstick test
- Asymptomatic Female Volunteers: These are subjects over the age of 18 who have no acute symptoms, volunteered to provide a urine sample, and are female.
  Interventions: Diagnostic Test: Urine dipstick test

INTERVENTIONS:
Diagnostic Test: Urine dipstick test — A sample of urine will be tested using a Mission Urinalysis Reagent Strip.

SUMMARY:
This is a prospective, observational study assessing the results of urine dipsticks on adult volunteers with no acute symptoms. We seek to determine the frequency of leukocytes or nitrites in this group of individuals.

DETAILED DESCRIPTION:
The urinalysis (UA) is one of the most commonly utilized tests in the emergency department (ED). In some busy EDs, a UA is routinely ordered by protocol on patients with abdominal pain, and in elderly patients, a UA is often ordered for a variety of chief complaints including dizziness and altered mental status. When these patients, who often do not specifically have symptoms of a urinary tract infection, have a urinalysis demonstrating pyuria or bacteria, it may be interpreted as an atypical presentation of a UTI. However, it is possible that these patients do not have urinary tract infections, but have baseline pyuria or bacteriuria. One prior study found that 5% of sexually active healthy women 18-40 have asymptomatic bacteriuria [1], and the rate of asymptomatic bacteriuria increases with age, such that it is present in 8-10% of women from 70-80 years of age [2]. Moreover, one prior article stated that 30-50% of residents of long term nursing facilities have positive urine cultures at any given time [3].

The above statistics come from the results of urine cultures. In the ED, the decision to treat or not treat a patient for a UTI is not made based upon culture results, but upon a urinalysis (microscopic or dipstick). Only one prior study has looked at the frequency of abnormal urinalyses in healthy individuals, and it found that over a third of asymptomatic women had at least 1+ leukocytes in their urine [4]. This is evidence that a substantial number of people who do not have symptomatic UTIs have UAs that could be interpreted as UTIs. If these results could be replicated and expanded to include a wider group of individuals (males, elderly patients, various races, etc.), it would provide valuable information about how we can better interpret and utilize the results of a UA.

Thus, the investigators propose a prospective study to assess the frequency of abnormal UAs in a wide variety of individuals without acute symptoms.

Urine samples will be obtained from adults with no acute symptoms, and performed urine dipsticks to assess the frequency of leukocytes or nitrites in the urine. Patients will be divided into groups to determine if there are certain factors (gender, age, or medical history) that increase the chance of having leukocytes or nitrites in the urine.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Able to spontaneously provide a urine sample

Exclusion Criteria:

* Any acute symptoms (including but not limited to vaginal bleeding, vaginal discharge, abdominal pain, back pain, dysuria, hematuria, and fever)
* Pregnancy
* Prisoner status
* Antibiotics within 72 hours
* Urologic procedure within a week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are all healthy volunteers, who are primarily family, friends, or acquaintances of study investigators.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Zitek, MD, Study Director — Nova Southeastern University
Locations (1):
- Kendall Regional Medical Center, Miami, Florida, United States

REFERENCES:
- [Background] Hooton TM, Scholes D, Stapleton AE, Roberts PL, Winter C, Gupta K, Samadpour M, Stamm WE. A prospective study of asymptomatic bacteriuria in sexually active young women. N Engl J Med. 2000 Oct 5;343(14):992-7. doi: 10.1056/NEJM200010053431402. PMID 11018165
- [Background] Kunin CM, McCormack RC. An epidemiologic study of bacteriuria and blood pressure among nuns and working women. N Engl J Med. 1968 Mar 21;278(12):635-42. doi: 10.1056/NEJM196803212781201. No abstract available. PMID 4866351
- [Background] Nicolle LE. Asymptomatic bacteriuria in institutionalized elderly people: evidence and practice. CMAJ. 2000 Aug 8;163(3):285-6. No abstract available. PMID 10951726
- [Background] Frazee BW, Enriquez K, Ng V, Alter H. Abnormal urinalysis results are common, regardless of specimen collection technique, in women without urinary tract infections. J Emerg Med. 2015 Jun;48(6):706-11. doi: 10.1016/j.jemermed.2015.02.020. Epub 2015 Apr 1. PMID 25841289

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Asymptomatic Male Volunteers | Asymptomatic Female Volunteers
Started | 96 | 104
Completed | 96 | 104
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asymptomatic Male Volunteers | Asymptomatic Female Volunteers | Total
Number analyzed (Participants) | 96 | 104 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (21.7) | 53.7 (23.6) | 50.1 (23.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 104 | 104
  Male | 96 | 0 | 96
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 86 | 96 | 182
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 96 | 104 | 200

OUTCOME MEASURES:

1. Primary Outcome: False Positive Urine
Description: A urine sample with at least 1+ leukocytes or positive nitrites on urine dipstick test will be considered a "false positive urine".
Time Frame: The urine is tested immediately, and results are available two minutes after placing the reagent strip in the urine.
Measure: Count of Participants; unit: Participants
Arm/Group | Asymptomatic Male Volunteers | Asymptomatic Female Volunteers
Number analyzed (Participants) | 96 | 104
Participants | 6 | 40

2. Secondary Outcome: Incidental Hematuria
Description: A urine sample with any blood on urine dipstick test will be considered to have "incidental hematuria"
Time Frame: The urine is tested immediately, and results are available two minutes after placing the reagent strip in the urine.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During urine specimen collection and survey completion (about 5 minutes)
Description: No adverse events were expected given the nature of the study.
Arm/Group | Asymptomatic Male Volunteers | Asymptomatic Female Volunteers
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/104
Other Adverse Events (participants affected / at risk) | 0/96 | 0/104

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/75/NCT04055675/Prot_SAP_000.pdf